CLINICAL TRIAL: NCT04793373
Title: Superiority of Epidural Placement Technique Using EpiFaith® Syringe Versus Conventional Glass Syringe in Laboring Paturients
Brief Title: Superiority of Epidural Placement Technique Using EpiFaith Syringe
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Protocol is being revised.
Sponsor: Harvard Medical School (HMS and HSDM) (Other)
Responsible Party: Principal Investigator, Jie Zhou, Assistant Professor, Harvard Medical School (HMS and HSDM)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2020P000677
Record Dates: First submitted 2021-03-09; First posted 2021-03-11 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: Anesthesia
MeSH Terms: interventions — Syringes

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- EpiFaith® group (Experimental): Study subject will have the epidural placement with an EpiFaith® syringe.
  Interventions: Device: Syringe
- Conventional group (Active Comparator): Study subject will have the epidural placement with a conventional glass syringe.
  Interventions: Device: Syringe

INTERVENTIONS:
Device: Syringe — A syringe will be used to detect the loss of resistance and needle's entry of epidural space.

SUMMARY:
The aim of this study is to evaluate the impact of EpiFaith® syringe on the establishment of successful epidural labor analgesia, change of elapsed time for identification of epidural space, and learning curve of CA-1 residents.

DETAILED DESCRIPTION:
We hypothesize that EpiFaith® syringe, in comparison with conventional glass syringe, will result in a similar overall success rate for catheter placement, but with a larger reduction in change of elapsed time for identification of epidural space and catheter placement of each practitioner. Moreover, we hypothesize that the cumulative learning summary curve using EpiFaith® syringe will be higher than conventional glass syringe in resident trainees, which will show the possible value of EpiFaith® syringe for teaching and learning obstetric epidural anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Females 18 years of age and older at screening
* Request labor epidural analgesia
* Able to give informed consent to participate in the study
* American Society of Anesthesiologists (ASA) class Ⅰ to Ⅲ health status
* BMI ≤ 40 kg/m2

Exclusion Criteria:

* BMI > 40 kg/m2; any contraindication to neuraxial anesthesia (coagulopathy, uncorrected hypovolemia, increased intracranial pressure, or local skin infection)
* Cardiac disease history, marked spinal deformity, previous spinal surgery, or impalpable anatomical landmarks
* Any allergy to bupivacaine or fentanyl

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Parturients who require labor epidural placement
Enrollment: 0 (Actual)
Dates: Start 2022-05-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Success of epidural localization | 30 minutes
  Defined as the catheter can be inserted into epidural space successfully; no occurence of inadvertent dural puncture

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States